CLINICAL TRIAL: NCT04977882
Title: Abdominal Drainage, Postoperative Antibiotico-prophylaxis and CME With D3 Lyphadenectomy Effect on Gastrointestinal Function in Laparoscopic Right Hemicolectomy With Intracorporeal Anastomosis for Right Colon Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Giuseppe Sigismondo Sica, Head of Minimally Invasive Surgery Unit, University of Rome Tor Vergata
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Registro sperimentazioni XX.21
Record Dates: First submitted 2021-07-15; First posted 2021-07-27 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Colon Cancer
Keywords: intracorporeal anastomosis; right hemicoletomy; colon cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients were initially randomized for postoperative management into three arms to receive prolonged antibiotic prophylaxis (ABX group), abdominal drain placement (DRAIN group) or neither (NONE group) (I level randomization). The same patients were further randomized for surgical technique in two arms to receive RRC (RRC group) or standard hemicolectomy with D2 dissection (STANDARD group) (II level of randomization).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Abdominal drainage (Experimental): 19 Fr abdominal drainage placed intraoperatevely in right paracolic gutter
  Interventions: Procedure: abdominal drainage; Procedure: Laparoscopic radical right colectomy with CME and D3 lymphadenectomy (RRC); Procedure: Laparoscopic standard D2 right hemicolectomy (STANDARD)
- Postoperative antibiotico-prophylaxis (Experimental): postoperative antibiotico-prophylaxis with Ceftriaxone 2gr and Metronidazole 1.5gr
  Interventions: Drug: Postoperative antibiotico-prophylaxis; Procedure: Laparoscopic radical right colectomy with CME and D3 lymphadenectomy (RRC); Procedure: Laparoscopic standard D2 right hemicolectomy (STANDARD)
- Control group (Sham Comparator): No drainage nor postoperative antibiotico-prophylaxis
  Interventions: Procedure: Laparoscopic radical right colectomy with CME and D3 lymphadenectomy (RRC); Procedure: Laparoscopic standard D2 right hemicolectomy (STANDARD)

INTERVENTIONS:
Procedure: abdominal drainage — 19 Fr abdominal drainage placed intraoperatively in right colic gutter
  Arms: Abdominal drainage
Drug: Postoperative antibiotico-prophylaxis — Ceftriaxone 2 gr and Metronidazole 1.5 gr per day for 2 days postoperatively
  Arms: Postoperative antibiotico-prophylaxis
Procedure: Laparoscopic radical right colectomy with CME and D3 lymphadenectomy (RRC) — the dissection starts over the landmark given by SMV. The SMV is freed anteriorly and on its right-hand side from all the lympho-adipose tissue. Once the SMV is fully exposed, the IC vessels are dissected and divided at the junction with the efferent vessels. The dissection moves upward along the same dissection line to identify the right colic vein and the GCTH. No medial to later dissection is carried out until the SMV is completely exposed before reaching the uncinate process of the pancreas. At this point the veins to the right colon are divided but gastroepiploic vein and artery are preserved unless the tumor is located at the hepatic flexure. The divided mesentery is lifted and tilted to the right, and the medial-to-later dissection starts following the embryological plane over Fredet's fascia. The mesocolon is divided on the right side of the middle colic artery and the right branches of the middle colic vessels are divided.
Procedure: Laparoscopic standard D2 right hemicolectomy (STANDARD) — A medial-to-lateral surgical dissection and high tie of the ileocolic vessels (IC) is undertaken without dissecting the anterior surface of the superior mesenteric vein (SMV). The gastro-colic trunk of Henle (GCTH) is not isolated and the right colic vein (when present) and the right branches of the middle colic vessels are taken more peripherical, during the division of the transverse mesocolon. The right gastroepiploic vessels are not dissected, nor divided, unless in proximity of the tumor

SUMMARY:
Monocentric, two-level factorial, parallel-arm, pilot randomized clinical trial, conducted comparing patients undergoing laparoscopic right hemicolectomy with ICA for right colon cancer in a single unit of a teaching hospital: Minimally Invasive Surgery Unit, Department of Surgical Sciences, Policlinico Tor Vergata, Rome, Italy.

ELIGIBILITY:
Inclusion Criteria:

* Right colon cancer
* Intracorporeal anastomosis
* Laparoscopic surgery
* Elective surgery
* informed consent signed

Exclusion Criteria:

* below 18 years old
* IBD
* ASA IV
* T4b
* Metastatic disease
* Preoperative steroids
* Conversion to open surgery
* Emergency surgery
* concomitant major operation
* preoperative infective status
* benign disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Tolerance to solid diet | 30 days postoperatively
  time to light diet tolerance

SECONDARY OUTCOMES:
White blood cell | 30 days postoperatively
  measured thousands/mL in I and III POD
Procalcitonine | 30 days postoperatively
  measured ng/ml in III and V POD
Days of hospitalization | 90 days postoperatively
  number of days of hospitalization
Readmission rate | 90 days postoperatively
  rate of hospital readmission
Mortality rate | 90 days postoperatively
  postoperative mortality
Surgical site infection rate | 30 days postoperatively
  postoperative wound infection
Anastomotic leak rate | 30 days postoperatively
  postoperative Ileocolic anastomotic leakage
Tolerance to liquid diet | 30 days postoperatively
  time to clear fluid tolerance
Time to first flatus | 30 days postoperatively
  Time to first flatus postoperatively
Time to first evacuation | 30 days postoperatively
  Time to first evacuation postoperatively
need of abdomen CTscan rate | 30 days postoperatively
  need of abdomen CTscan
C-Reactive Proteine | 30 days postoperatively
  measured mg/L in I and III POD

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rome Tor Vergata, Rome, Italy

REFERENCES:
- [Derived] Sica GS, Siragusa L, Pirozzi BM, Sorge R, Baldini G, Fiorani C, Guida AM, Bellato V, Franceschilli M. Gastrointestinal functions after laparoscopic right colectomy with intracorporeal anastomosis: a pilot randomized clinical trial on effects of abdominal drain, prolonged antibiotic prophylaxis, and D3 lymphadenectomy with complete mesocolic excision. Int J Colorectal Dis. 2024 Jul 6;39(1):102. doi: 10.1007/s00384-024-04657-0. PMID 38970713